CLINICAL TRIAL: NCT05792150
Title: Real World Data and Long-term FU of Pre-/Perimenopausal Women With Luminal EBC With Intermediate to High Clinical and Low Genomic Recurrence-risk Measured by MammaPrint®, Treated by SOC ET+OFS or SOC Chemotherapy Treatment Followed by ET
Brief Title: PROOFS-Registry - Premenopausal Women With Breast Cancer Optimally Treated With OFS
Acronym: PROOFS
Status: Recruiting | Type: Observational
Sponsor: West German Study Group (Other)
Collaborators: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: WSG-NIS04 / PROOFS
Record Dates: First submitted 2023-02-13; First posted 2023-03-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Female Breast Cancer
Keywords: HR+; HER2-; EBC; early breast cancer; female; OFS; ET; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is only limited data for premenopausal patients in general, as well as for differences in the use of OFS in the subgroups of pre- and perimenopausal patients, respectively. The WSG ADAPT trial data on the impact of postmenopausal status and/or use of OFS within 3-4 weeks endocrine induction therapy show relevant impact of OFS/postmenopausal status on Ki-67 response; also, secondary amenorrhea after (neo-)adjuvant chemotherapy was a positive predictor of outcome due to OFS [8, 9].

This registry will give insights in the real-world use of OFS and the effect of secondary amenorrhea in female pre- and perimenopausal patients with or without previous use of chemotherapy and with different endocrine treatments (ET +/- GnRH).

As adherence over time (5-10 years) plays a major role in the endocrine treatment, the registry will follow patients' treatments for up to 10 years and include QoL information.

Results of MammaPrint® (MammaPrint® Index) as indicating factor for chemotherapy use and risk classification, thus, choice of adjuvant treatment (chemotherapy, OFS combined with endocrine therapy, or endocrine therapy alone) will be correlated to outcome under real-world conditions.

Baseline, treatment, and relapse data shall be collected to gain further insight in the treatment paths, treatment adherence, and outcome of such patients.

DETAILED DESCRIPTION:
This registry aims

* to confirm an excellent outcome in pre-/perimenopausal patients treated by endocrine therapy (+ ovarian suppression) in patients with low genomic risk by MammaPrint® without chemotherapy use in a real-world setting.
* to evaluate management of ovarian function in patients treated by adjuvant chemotherapy according to investigator decision.
* to evaluate adherence to endocrine therapy (+/- ovarian function suppression).
* to evaluate the prognostic impact of clinicopathological markers (e.g., estrogen receptor (ER), progesterone receptor (PR), HER2 receptor, Ki-67 at baseline and after preoperative endocrine therapy (if any performed) by local pathology assessment compared to genomic signature result.
* to assess the course of quality of life (QLQ BR23 and QLQ-C30) until 5 years of treatment with OFS (Baseline, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, 5 years)

In general, WSG aim to assess the quality of surveillance care in younger breast cancer patients. WSG want to gain knowledge about endocrine induction treatment for indication of chemotherapy followed by endocrine treatment or endocrine treatment alone. Also, WSG aim at changes in duration of endocrine treatment (especially in high-risk patients up to 10 years) and introduction of intensified endocrine therapy (OFS) in combination with GnRH-analogues since publication of the SOFT and TEXT trials.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for participation in the registry only if they meet all the following criteria:

* Female breast cancer patients
* Pre- or perimenopausal at registry entry (age <60 years and state after hysterectomy or amenorrhea for <12 months; confirmation by blood hormone levels (FSH and estradiol in premenopausal range as per local normal range) recommended)
* Primary tumor diagnosis not older than three months prior to inclusion (primary diagnosis defined as date of initial tumor biopsy)
* Estrogen- and/or progesterone-receptor-positive/HER2 negative early breast cancer without any clinical signs of metastases
* Adequate risk for recurrence:
* intermediate clinical risk for recurrence, defined as (clinical in case of neoadjuvant treatment):
* c/pT1 and
* c/pN0 and
* Ki-67 15-24% or
* G2 or
* patients, who do not meet these criteria but are at intermediate clinical risk for recurrence at investigator decision (e.g., very young age, low expression of hormone receptors, existing co-morbidities, familial cancer burden, etc.) can be included on individual decision basis or
* high clinical risk for recurrence, defined as either (clinical in case of neoadjuvant treatment):
* c/pT2-4 or
* c/pN1 or
* Ki-67 ≥25% or
* G3
* Low genomic risk of recurrence by MammaPrint® (tested on treatment naïve tumor specimen)
* Luminal-type by BluePrint®
* Treatment according to standard-of-care (e.g., AGO Guidelines) planned or started (until completion of local therapy the latest (including started or completed endocrine induction therapy), started, or planned adjuvant or neoadjuvant treatment)
* Availability of untreated tumor material (core biopsy if preoperative endocrine therapy performed or neoadjuvant treatment intended or surgery specimen)
* Capability to give written informed consent
* Nodal positive patients will be accepted to the registry up to 25% of the genomic low/ultralow-risk population (n=441).

Exclusion Criteria:

Patients will not be eligible for the registry for any of the following reasons:

* Any other genomic testing, besides MammaPrint®, has been performed on the tumor material
* Medical or psychological conditions that would not permit the patient to sign informed consent
* Legal incapacity or limited legal capacity
* Current participation in any interventional clinical trial which tests anticancer drugs, immunotherapeutics, or antibody treatment for any type of neoplasm
* Non-compliance of the patient

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: For this registry, it is planned to screen N=3000 pre- and perimenopausal patients with early breast cancer who meet the inclusion criteria, i.e., intermediate to high clinical risk for recurrence, and who will receive or have received a routine genomic testing by MammaPrint® with a low/ultralow genomic risk.
  It is anticipated that 75% of these patients will be nodal negative and 25% nodal positive.
Sampling Method: Non-Probability Sample
Enrollment: 1470 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2035-03 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
5-year distant recurrence-free interval (dRFI, according to STEEP criteria version 2.0) | 5 years
  dRFIin all patients treated by (intensified) endocrine therapy alone (and with ovarian suppression in cases with enhanced clinical risk according to current AGO-recommendations)

SECONDARY OUTCOMES:
10-year dRFI | 10 years
  dRFI, according to STEEP criteria 2.0, in all patients treated by (intensified) endocrine therapy alone (with ovarian suppression in cases with higher clinical risk)
5-year dRFI | 5 years
  dRFI, according to STEEP criteria 2.0,in all patients treated by SOC chemotherapy treatment followed by ET+/-OFS
10-year dRFI | 10 years
  dRFI, according to STEEP criteria 2.0,in all patients treated by SOC chemotherapy treatment followed by ET+/-OFS
5-year dDFS | 5 years
  distant disease-free survival (dDFS, according to STEEP 2.0) in all patients and all treatment groups (i.e., patients treated by ET alone, ET + GnRH, chemotherapy followed by ET, chemotherapy followed by ET + GnRH, OFS-treated patients)
10-year dDFS | 10 years
  distant disease-free survival (dDFS, according to STEEP 2.0) in all patients and all treatment groups (i.e., patients treated by ET alone, ET + GnRH, chemotherapy followed by ET, chemotherapy followed by ET + GnRH, OFS-treated patients)treatment followed by ET+/-OFS
5-year OS | 5 years
  overall survival (OS) in all patients and all treatment groups
10-year OS | 10 years
  overall survival (OS) in all patients and all treatment groups
5-year breast cancer-free interval (BCFI, according to STEEP 2.0) | 5 years
  BCFI in all patients and all treatment groups
10-year breast cancer-free interval (BCFI, according to STEEP 2.0) | 10 years
  BCFI in all patients and all treatment groups
EORTC quality of life questionnaire BR23 | every 3 months within 1st year
  compare the course of Qol between baseline and further defined timepoints; 23 items, symptom scales/items and functional scales/items, all of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
EORTC quality of life questionnaire C30 | every 3 months within 1st year
  compare the course of Qol between baseline and further defined timepoints; 30 items, 10 subscales, the higher the rating, the worse.
EORTC quality of life questionnaire BR23 | every 6 months within 2nd year
  compare the course of Qol between baseline and further defined timepoints; 23 items, symptom scales/items and functional scales/items, all of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
EORTC quality of life questionnaire C30 | every 6 months within 2nd year
  compare the course of Qol between baseline and further defined timepoints; 30 items, 10 subscales, the higher the rating, the worse.
EORTC quality of life questionnaire BR23 | yearly until 5 years
  compare the course of Qol between baseline and further defined timepoints; 23 items, symptom scales/items and functional scales/items, all of the scales and single-item measures range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, whilst a high score for the symptom scales represents a high level of symptomatology or problems.
EORTC quality of life questionnaire C30 | yearly until 5 years
  compare the course of Qol between baseline and further defined timepoints; 30 items, 10 subscales, the higher the rating, the worse.
adherence to OFS and endocrine treatment | 10 years
  Duration of intake of OFS and endocrine treatment in all patients
concordance between BluePrint®/MammaPrint® molecular subtyping results vs. pathological immune-histochemistry results | 10 years
  concordance between BluePrint®/MammaPrint® molecular subtyping results and pathological immune-histochemistry results with respect to tumour type
endocrine response measured by post-endocrine Ki-67 | 10 years
  post-endocrine Ki-67 (≤10% and/or relative change vs. baseline) in patients treated by preoperative ET
5-year iDFS in node-negative patients with ultralow MammaPrint | 5 years
  node-negative patients with ultralow MammaPrint® treated by shorter duration of ET (2-3 years at investigator decision)
10-year iDFS in node-negative patients with ultralow MammaPrint | 10 years
  node-negative patients with ultralow MammaPrint® treated by shorter duration of ET (2-3 years at investigator decision)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Gluz, PD Dr., Principal Investigator — Westdeutsche Studiengruppe GmbH; Rachel Wuerstlein, Prof. Dr., Principal Investigator — Westdeutsche Studiengruppe GmbH; Monika Graeser, PD Dr., Study Director — Westdeutsche Studiengruppe GmbH; Nadia Harbeck, Prof. Dr., Principal Investigator — LMU Clinics, Breast Centre and CCC; Sherko Kuemmel, Prof. Dr., Principal Investigator — KEM, Clinics Essen-Mitte; Ulrike Nitz, Prof. Dr., Study Director — Westdeutsche Studiengruppe GmbH; Andreas Hartkopf, Prof. Dr., Principal Investigator — Univewrsity Hospital Tuebingen
Locations (71):
- Germany (71):
  - Klinikum-Mittelbaden GmbH, Studienzentrale/Brustzentrum, Baden-Baden, Baden-Wurttemberg
  - Helios Klinikum Pforzheim, Brustzentrum, Pforzheim, Baden-Wurttemberg
  - Diakonieklinikum Stuttgart, Brustzetrum, Stuttgart, Baden-Wurttemberg
  - Universitätsfrauenklinik Ulm - Frauenheilkunde und Geburtshilfe, Ulm, Baden-Wurttemberg
  - GRN Klinik Weinheim/ Gynäkologie/Brustzentrum, Weinheim, Baden-Wurttemberg
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe, Baden-Wüttemberg
  - Studienzentrum Onkologie Ravensburg, Ravensburg, Baden-Wüttemberg
  - Klinikum St. Marien Amberg, Amberg, Bavaria
  - HOP Gemeinschaftspraxis Dres. Heinrich/Bangerter, Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Augsburg, Brustzentrum, Augsburg, Bavaria
  - Medias Klinikum, Burghausen, Bavaria
  - Klinikum Fürstenfeldbruck, Westdeutsches Brust- Centrum, Fürstenfeldbruck, Bavaria
  - Klinikum der Universität München, München, Bavaria
  - Med. Zentrum f. Hämatologie und Onkologie München, München, Bavaria
  - Caritas-Krankenhaus St. Josef, Klinik für Frauenheilkunde & Geburtshilfe, Regensburg, Bavaria
  - Gemeinschaftskrankenhaus/ Brustzentrum Havelhöhe, Berlin, Brandenburg
  - Klinikum Luckenwalde, Luckenwalde, Brandenburg
  - Klinikum Bremerhaven Reinkenheide, Bremerhaven, City state Bremen
  - Gesundheitszentrum Wetterau gGmbH Hochwaldkrankenhaus Bad Nauheim, Bad Nauheim, Hesse
  - Gynäkologische- Geburtshilfliche Klinik, Bad Soden am Taunus, Hesse
  - Klinikum Hanau GmbH, Hanau, Hesse
  - Elisabethkrankenhaus Kassel, Brustzentrum, Kassel, Hesse
  - Universität Marburg, Klinik für Frauenheilkunde, Brustzentrum, Marburg, Hesse
  - St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden, Hesse
  - DIAKOVERE Henriettenstift, Hanover, Lower Saxony
  - Ärztehaus am Bahnhofsplatz, Hildesheim, Lower Saxony
  - Studienzentrum Untere Ems, Leer, Lower Saxony
  - Onkologische Praxis Oldenburg, Gemeinschaftspraxis für Innere Medizin, Hämatologie und Onkologie, Oldenburg, Lower Saxony
  - Klinikum Südstadt, Rostock, Mecklenburg-Vorpommern
  - Marienhospital Aachen, Aachen, North Rhine-Westphalia
  - Gynäkologisches Zentrum, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Bonn Frauenheilkunde, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Senologie, Bonn, North Rhine-Westphalia
  - Kliniken der Stadt Köln, Cologne, North Rhine-Westphalia
  - St. Vincenz-Krankenhaus Datteln, Datteln, North Rhine-Westphalia
  - Klinikum Dortmund gGmbH, Beurhausstr.40, Dortmund, North Rhine-Westphalia
  - Evangelisches Krankenhaus BETHESDA zu Duisburg GmbH, Brustzentrum, Duisburg, North Rhine-Westphalia
  - Luisenkrankenhaus GmbH Co KG, Düsseldorf, North Rhine-Westphalia
  - Marien Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Evang. Kliniken Essen Mitte, Interdisziplinäres Brustkrebszentrum, Essen, North Rhine-Westphalia
  - St. Antonius Hospital Kleve (Katholisches Kral Leistner Zentrum), Goch, North Rhine-Westphalia
  - AGAPLESION Allgemeines Krankenhaus Hagen, Hagen, North Rhine-Westphalia
  - St. Barbara Klinik, Hamm, North Rhine-Westphalia
  - Gemeinschaftskrankenhaus Herdecke gemeinnützige GmbH, Herdecke, North Rhine-Westphalia
  - Klinikum Leverkusen, Am Gesundheitspark, Leverkusen, North Rhine-Westphalia
  - Katholisches Klinikum Lünen/Werne, Lünen, North Rhine-Westphalia
  - Brustzentrum Niederrhein, Johanniter Bethesda Krankenhaus, Mönchengladbach, North Rhine-Westphalia
  - St. Franziskus-Hospital, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Frauenklinik St. Louise - St. Vincenz-Krankenhaus GmbH, Paderborn, North Rhine-Westphalia
  - Mathias-Spital-Rheine, Rheine, North Rhine-Westphalia
  - Praxisnetzwerk Hämatologie/int. Onkologie, Troisdorf, North Rhine-Westphalia
  - Christliches Klinikum Unna gGmbH, Unna, North Rhine-Westphalia
  - Evangelisches Krankenhaus Wesel GmbH, Wesel, North Rhine-Westphalia
  - Helios Klinikum Wuppertal, Wuppertal, North Rhine-Westphalia
  - Klinikum Worms, Worms, Rhineland-Palatinate
  - Krankenhaus St. Elisabeth und St. Barbara Halle/Saale, Halle, Saxony-Anhalt
  - Altmark- Klinikum, Salzwedel, Saxony-Anhalt
  - Medionko - Praxisklinik Krebsheilkunde Frauen, Berlin
  - St. Gertrauden Krankenhaus Brustzentrum City Berlin, Berlin
  - DRK Kliniken Berlin Köpenick, Berlin
  - Marienhospital, Klinik für Gynäkologie und Geburtshilfe, Bottrop
  - Hämatologie/Onkologie Praxis, Bremen
  - DIAKO Ev. Diakonie-Krankenhaus gemeinnützige GmbH, Bremen
  - Universitätsklinikum Erlangen, Erlangen
  - AGAPLESION Diakonie Hamburg, Hamburg
  - Gynäkologische Praxisklinik Hamburg-Harburg, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Helios Klinikum Krefeld, Zentrum für Ambulante Gynäkologische Onkologie - Studienabteilung, Krefeld
  - MKS St. Paulus Schwerte (ehemals Marienkrankenhaus), Schwerte
  - Klinikum Traunstein, Frauenklinik Südostbayern, Traunstein

IPD SHARING:
Plan to Share IPD: No